CLINICAL TRIAL: NCT03076905
Title: F901318 - A Phase I, Single Intravenous Dose, Safety, Tolerability and Pharmacokinetics Study in Healthy Male and Female Subjects
Brief Title: Pharmacokinetics of IV Formulation
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: study no longer required in current format
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F901318-01-10-17; QCL117986 (Other: Quotient Clinical)
Record Dates: First submitted 2017-03-06; First posted 2017-03-10 (Actual); Last update posted 2017-11-01 (Actual); Status verified 2017-03

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — olorofim

STUDY DESIGN:
Intervention Model Description: Assessment of IV pharmacokinetics
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IV drug (Experimental): AUC0-t of single intravenous dose of F901318
  Interventions: Drug: F901318

INTERVENTIONS:
Drug: F901318 — Evaluation of AUC0-t

SUMMARY:
Open label evaluation of a single intravenous dose of F901318 to healthy male and female subjects with pharmacokinetic and safety and tolerability evaluation.

DETAILED DESCRIPTION:
Open label single intravenous dose, single group study. Eight subjects (ideally 4 male and 4 female, minimum of two females) will be studied. The drug product will be a F901318 solution for infusion (6mg/mL). The dose will be 4 mg/kg delivered in the fasted state (8 hours minimum) by intravenous infusion over 2 hours. Each subject will be on study for approximately 6 weeks. Each subject will reside at the Clinical Research Unit (CRU) from Day -1 (the day before dosing) to Day 4 (72 hours post-dose). Blood samples for pharmacokinetic evaluation will be obtained up to and including 120 hours post dose. Safety and tolerability will also be assessed.

Subjects will return to the clinical unit at 96 and 120 hours for pharmacokinetic blood sampling.

All subjects will return for a post-study visit 8 to 10 days after the dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males or females of any ethnic origin between 18 and 55 years or age and weighing between 50 and 100kg.
2. Females of child bearing potential must be established on a reliable form of contraception and have a negative pregnancy test at screening and Day -1
3. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (hepatic transaminases must be within normal limits, congenital non haemolytic hyperbilirubinaemia is acceptable)
4. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions

Exclusion Criteria:

1. Female and male subjects who are not, or whose partners are not willing to use appropriate contraception with two reliable forms of contraception or who are not otherwise unable to conceive children (hysterectomy, oophorectomy, tubal ligation or post menopausal).
2. Subjects who have received any prescribed systemic or topical medication within 14 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety
3. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the dose administration (with the exception of vitamin/mineral supplements and paracetamol) unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic profile (AUC0-t) | 120 hours
  AUC0-t

SECONDARY OUTCOMES:
Tolerability (Adverse events) | 120 hours
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Litza McKenzie, MD, Principal Investigator — Quotient Clinical

IPD SHARING:
Plan to Share IPD: No